CLINICAL TRIAL: NCT05304507
Title: Tailored Model for Implementation of Injury Prevention Training in Youth Handball Compared With Current Practice: A Pilot Study of the I-PROTECT Model
Brief Title: Pilot Study of a Tailored Model for Implementation of Injury Prevention Training in Youth Handball (the I-PROTECT Model)
Acronym: I-PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-02952; 2014/713 (Other: Regional Ethical Review Board in Lund, Sweden)
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Non-randomized pilot study
Who Masked: Outcomes Assessor
Masking Description: An independent statistician, blinded to group allocation, will analyze data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PROTECT model (Experimental): The I-PROTECT model is an end-user-driven intervention including evidence-based, theory-informed, and context-specific injury prevention training for youth handball, and an associated implementation strategy.
  Interventions: Behavioral: I-PROTECT model
- Control group (Active Comparator): Youth coaches in the control group club will be asked to use injury prevention training available in the coach education material ("Ready for handball"), i.e., current practice in Sweden.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: I-PROTECT model — The I-PROTECT model is based on existing research and knowledge of experts in sport medicine, sport psychology and implementation science, with the involvement of end-users throughout the process. The interdisciplinary intervention includes exercises based on physical and psychological principles of effective injury prevention training, specifically tailored for youth handball players, and support for developing a continuous implementation strategy. The intervention is delivered through a mobile application specifically developed for the I-PROTECT project (the I-PROTECT GO), including coach, player, club administrator, and caregiver modules. Coaches are introduced to the intervention in a workshop, and they will conduct the exercises with their teams during handball practice. Players will have support for conducting exercises on their own, and club administrators for developing an implementation strategy. Caregivers will have tailored information about injury prevention training.
  Arms: I-PROTECT model
Behavioral: Control group — Youth coaches in the control group club will be asked to use injury prevention training available in the coach education material ("Ready for handball"), i.e., current practice in Sweden.
  Arms: Control group

SUMMARY:
This pilot study aims to test a tailored model (the I-PROTECT model) for implementation of injury prevention training in youth handball compared with current practice.

DETAILED DESCRIPTION:
Injury prevention training is effective in reducing musculoskeletal injuries in youth athletes but has had limited public health impact because it is not widely or properly implemented. The lack of involving end-users at the individual and organizational levels is a main contributor to insufficient implementation.

This is a non-randomized pilot study included in the "Implementing injury Prevention training ROutines in TEams and Clubs in youth Team handball (I-PROTECT)" project. The overall aim of I-PROTECT is to achieve wide-spread, sustained and high-fidelity use of evidence-based injury prevention training in youth handball through behavior change at multiple levels within the sports delivery system (individual and organizational levels). The I-PROTECT model is evidence-based, theory-informed, and context-specific injury prevention training specifically tailored for youth handball players, incorporating physical and psychological components and an associated implementation strategy. The process of developing the I-PROTECT model has been described.

In a prospective single-case study (ClinicalTrials.gov registration number: NCT04481958), the I-PROTECT model was implemented and tested in all youth teams (n=19) of two clubs during the 2020/2021 handball season. Due to Covid pandemic restrictions, handball training was only performed for about 2 months, thus, affecting intervention implementation and data collection. To further evaluate, develop, and finalize the I-PROTECT model, we will in the current study conduct pilot testing in clubs not involved in developing the model, before testing the model in a larger scale study.

Two clubs in Sweden offering handball for youth players will be recruited by convenience sampling. One club will use the I-PROTECT model (experimental) and one club will use current practice (control). Intervention will be approx. 6 weeks. Data will be collected among stakeholders (players, coaches, club administrators, caregivers) before, during and after the intervention. Parametric, or non-parametric, tests will be used as appropriate for main and secondary outcomes. Data will be used to calculate sample size in the main outcome for a larger scale study as well as to assess implementation determinants.

ELIGIBILITY:
Stakeholders (players, coaches, caregivers, club administrators) of all youth teams (13-17 years) in two community handball clubs will be eligible for participation.

Inclusion Criteria:

* Players: ages 13-17 years and training ≥2 times/week in a team
* Coaches: leading ≥1 training session/week
* Caregivers: directly associated with the eligible players
* Club administrators: engagement in the issues of sports injury, coach education or policy development for youth players

Exclusion Criteria:

* Employed/paid players
* Stakeholder other than the groups listed in inclusion criteria

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of injury prevention training | Study start up to end of study (6 weeks)
  Frequency of injury prevention training on a team level, reported by coaches weekly (0, 1, 2, 3 or more session/week). Using injury prevention training for two session or more per week at regular handball training over the intervention period will signify that injury prevention is implemented in a team (binary outcome: ≥2 per week or <2 per week).

SECONDARY OUTCOMES:
Adoption and fidelity (coaches) | Study start up to end of study (6 weeks)
  Coaches' weekly report if they have followed the program as intended.
Implementation determinants | Baseline
  Questionnaire data for implementation determinants will be collected for coaches and caregivers. Questions aligned with the Health Action Process Approach (HAPA) theory and the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework will be adapted to each stakeholder group.
Implementation determinants | After study end at approx. 6 weeks
  Questionnaire or interview data for implementation determinants will be collected for all stakeholders (players, coaches, caregivers, club representatives). Questions aligned with the Health Action Process Approach (HAPA) theory and the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework will be adapted to each stakeholder group. Data will also be gathered (e.g., focus groups interviews) to enable an in-depth understanding of potential barriers and facilitators, acceptability, usability, and sustainability of the I-PROTECT model, including its packaging, and of potential barriers for filling in questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Prof, Principal Investigator — Lund University
Locations (1):
- Eva Ageberg, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Share published data on reasonable request

REFERENCES:
- [Background] Ageberg E, Bunke S, Nilsen P, Donaldson A. Planning injury prevention training for youth handball players: application of the generalisable six-step intervention development process. Inj Prev. 2020 Apr;26(2):164-169. doi: 10.1136/injuryprev-2019-043468. Epub 2020 Feb 4. PMID 32019772